CLINICAL TRIAL: NCT03369938
Title: Exercise Training in Patients With Left Ventricular Assist Device
Acronym: Ex-VAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); University of Göttingen (Other); University Medicine Greifswald (Other); Technical University of Munich (Other); University of Leipzig (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Frank Edelmann, Professor for Cardiovascular Prevention and Clinical Heart Failure Research, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ex-VAD
Record Dates: First submitted 2017-11-15; First posted 2017-12-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: left ventricular assist device; exercise training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise training intervention (Experimental)
  Interventions: Other: exercise training intervention
- usual care (No Intervention)

INTERVENTIONS:
Other: exercise training intervention — structured aerobic endurance/resistance training on top of usual care for 12 weeks (3x/week)
  Arms: exercise training intervention

SUMMARY:
The objective of the study is to test whether 12 weeks of structured supervised exercise training on top of usual care improves functional capacity in patients with end-stage heart failure with continuous flow left ventricular assist device (LVAD).

ELIGIBILITY:
Inclusion Criteria:

* chronic end-stage systolic heart failure
* stable on left ventricular assist device, meaning

  1. no major change in therapeutic regime within past 4 weeks: no new additional disease modifying drug (ACE inhibitor, ARB, sacubitril, beta-blocker), no change in disease modifying drug dosage more than 50% (excluded: diuretics), no initiation of a cardiac rehabilitation for a minimum of 4 weeks
  2. post implantation ≥ 3 months
  3. expected further period on the device for a minimum of 3 months after recruitment into the study
* ability to complete the study in compliance with the protocol.
* general ability of the patient to declare willingness to participate in the trial.
* written informed consent

Exclusion Criteria:

* acute illness that does not allow exercise, including unstable heart failure, acute myocarditis, acute pericarditis, stroke
* untreated life-threatening cardiac arrhythmias
* uncontrolled hypertension
* intracardiac thrombus
* inability to perform cardiopulmonary exercise testing at least 1 minute at 20W
* uncontrolled diabetes
* uncontrolled kidney disease
* recent embolism
* concurrent, continuous, or intermittent dobutamine therapy
* complex ventricular arrhythmia at rest or appearing with exertion
* supine resting heart rate > 100 beats per minute
* severe pulmonary instability
* hemodynamically relevant valvular disorders
* significant change in cardiovascular medication within the previous 4 weeks (see inclusion criteria)
* severe anemia (hemoglobin <8 g/dl), however patients with moderate anemia (hemoglobin <11 g/dl) may be recruited if clinically stable (investigator assessment)
* clinically relevant musculoskeletal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change in maximal exercise capacity | after 12 weeks of treatment
  cardiopulmonary exercise testing (CPET; peakVO2)

SECONDARY OUTCOMES:
change in ventilatory efficacy | after 12 weeks of treatment and 12 weeks of follow-up
  cardiopulmonary exercise testing (CPET; VE/VCO2 slope)
change in submaximal exercise tolerance | after 12 weeks of treatment and 12 weeks of follow-up
  6-minute-walk distance (m), anaerobic threshold (VO2 at AT)
change in muscle strength | after 12 weeks of treatment and 12 weeks of follow-up
  handgrip (kg)
change in body composition | after 12 weeks of treatment and 12 weeks of follow-up
  % fat mass
Kansas City Cardiomyopathy Questionnaire (KCCQ) | after 12 weeks of treatment and 12 weeks of follow-up
  patient-reported measure of quality of life for patients with heart failure
36-Item Short Form Survey (SF-36) | after 12 weeks of treatment and 12 weeks of follow-up
  patient-reported measure of health status
Patient Health Questionnaire (PHQ-9) | after 12 weeks of treatment and 12 weeks of follow-up
  patient-reported measure of presence and severity of depression
change in echocardiographic parameters of cardiac morphology and function at rest and during exercise | after 12 weeks of treatment and 12 weeks of follow-up
  left ventricular ejection fraction (%)
change in echocardiographic parameters of cardiac morphology and function at rest and during exercise | after 12 weeks of treatment and 12 weeks of follow-up
  left ventricular end diastolic volume (ml)
change in echocardiographic parameters of cardiac morphology and function at rest and during exercise | after 12 weeks of treatment and 12 weeks of follow-up
  left ventricular end diastolic diameters (mm)
change in echocardiographic parameters of cardiac morphology and function at rest and during exercise | after 12 weeks of treatment and 12 weeks of follow-up
  tricuspid annular plane systolic excursion (TAPSE; mm)
change in markers of neuroendocrine activation | after 12 weeks of treatment and 12 weeks of follow-up
  NT-proBNP (ng/l)
change in daily physical activity | up to 12 weeks of treatment and 12 weeks of follow-up
  physical activity diary
change in daily physical activity | up to 12 weeks of treatment and 12 weeks of follow-up
  accelerometry

OTHER OUTCOMES:
adherence to exercise training | up to 12 weeks of treatment
  accelerometry

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Charité - Universitätsmedizin Berlin und Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universität München und Klinikum der Universität München, München

REFERENCES:
- See also: Ex-VAD trial website — http://ex-vad.dzhk.de/